CLINICAL TRIAL: NCT02263976
Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Rising Inhaled BEA 2180 BR Doses (2.5 μg to 1600 μg Cation Administered With the Respimat®) in Healthy Male Subjects, Alone and Followed by Methacholine Challenge. A Randomised, Double-blind Within Dose Group, Placebo-controlled Study, With a 36 μg Tiotropium Bromide Single Dose Sub-study (Open, Two-fold Crossover).
Brief Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of BEA 2180 BR in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.1; 1205.9001 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Methacholine Chloride; Tiotropium Bromide

ARMS (3):
- BEA 2180 BR (Experimental): single rising doses
  Interventions: Drug: BEA 2180 BR; Device: Respimat® A 4; Drug: Methacholine Chloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Respimat® A 4; Drug: Methacholine Chloride
- Sub-Study (Experimental)
  Interventions: Drug: Methacholine Chloride; Drug: Spiriva

INTERVENTIONS:
Drug: BEA 2180 BR
  Arms: BEA 2180 BR
Drug: Placebo
  Arms: Placebo
Device: Respimat® A 4
  Arms: BEA 2180 BR; Placebo
Drug: Methacholine Chloride — methacholine challenge test
Drug: Spiriva
  Other Names: tiotropium bromide
  Arms: Sub-Study

SUMMARY:
Main study: To investigate safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of BEA 2180 BR Sub-study; To investigate whether treatment with 36 μg tiotropium bromide is able to protect of methacholine-induced bronchoconstriction compared to baseline (methacholine challenge at screening).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory test
* No finding deviating from normal and of clinical relevance
* No evidence of a clinically relevant concomitant disease
* Age ≥ 30 and Age ≤ 55 years
* Body Mass Index (BMI) ≥ 18.5 and BMI < 30 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator (or his deputy)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance

Exclusion criteria specific for this study:

* Bronchial hyperreactivity as demonstrated by a 45% change of SGaw at or below a cumulative methacholine concentration of 10 mg/mL = 1%
* Asthma or bronchial hyperreactivity
* Allergic rhinitis (hay fever)
* Glaucoma
* Urinary tract obstruction
* Epilepsy
* History of cardiovascular disease
* History of peptic ulcer disease
* History of thyroid disease

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2003-08; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically significant changes in vital signs | up to 14 days after last drug administration
  blood pressure, pulse rate, respiratory rate, oral body temperature
Number of subjects with clinically significant changes in laboratory parameters | up to 14 days after last drug administration
Changes from baseline in airway resistance (Raw) | up to 120 hours after drug administration
  assessed by body plethysmography
Changes from baseline in specific airway conductance (sGaw) | up to 120 hours after drug administration
  assessed by body plethysmography
Number of subjects with clinically significant findings in 12-lead ECG (electrocardiogram) | up to 14 days after last drug administration
Number of subjects with adverse events | up to 14 days after last drug administration
Assessment of tolerability by investigator on a 5-point scale | within 14 days after last drug administration

SECONDARY OUTCOMES:
Changes from baseline in salivary secretion | up to 24 hours after drug administration
Changes from baseline in pupil diameter of each eye | up to 4 hours after drug administration
  pupillometry
Maximum measured concentration of the analyte in plasma (Cmax) | up to 240 hours after drug administration
Measured concentration of the analyte in plasma (C) for several time points | up to 24 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 240 hours after drug administration
Amount of parent drug that is eliminated in urine (Ae) | up to 312 hours after drug administration
Fraction of administered drug excreted unchanged in urine (fe) | up to 312 hours after drug administration
Area under the concentration-time curve of the analyte in plasma (AUC) | up to 240 hours after drug administration
Renal clearance of the analyte (CLR) | up to 312 hours after drug administration
Terminal rate constant of the analyte in plasma (λZ) | up to 240 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 240 hours after drug administration
Mean residence time of the analyte in the body after inhaled administration (MRTinh) | up to 240 hours after drug administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | up to 240 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (VZ/F) | up to 240 hours after drug administration